CLINICAL TRIAL: NCT02445612
Title: Long Term Follow Up to a Phase I/II, Open-Label, Multi-Center, Prospective Study to Determine the Safety and Tolerability of Sub-retinal Transplantation of Human Embryonic Stem Cell Derived Retinal Pigmented Epithelial (MA09-hRPE) Cells in Patients With Stargardt's Macular Dystrophy (SMD)
Brief Title: Long Term Follow Up of Sub-retinal Transplantation of hESC Derived RPE Cells in Stargardt Macular Dystrophy Patients
Status: Completed | Type: Observational
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 7316-CL-0004; ACT MA09-hRPE 001(SMD)LTFU (Other: Sponsor)
Record Dates: First submitted 2015-05-13; First posted 2015-05-15 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Stargardt's Macular Dystrophy
Keywords: fundus flavimaculatus; ASP7316; SMD; long term follow-up; juvenile macular dystrophy
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Experimental: MA09-hRPE: Sub-retinal transplantation of MA09-hRPE cells
  Interventions: Biological: MA09-hRPE

INTERVENTIONS:
Biological: MA09-hRPE — Cohort 1 50,000 cells Cohort 2 100,000 cells Cohort 2a Better Vision 100,000 cells Cohort 3 150,000 cells Cohort 4 200,000 cells
  Other Names: ASP7316

SUMMARY:
The purpose of this study is to evaluate the long term safety and tolerability of MA09-hRPE cellular therapy in patients with advanced Stargardt's Macular Dystrophy (SMD) from one to five years following the surgical procedure to implant the MA09-hRPE cells.

DETAILED DESCRIPTION:
This study is a long term, follow up to the ACT MA09-hRPE 001 phase I/II trial, the phase I/II trial (referred to as the core protocol) was an open-label, non-randomized, dose escalation, multi-center trial. Thirteen SMD patients were treated in this trial. Ten patients with profound vision loss (visual acuity <=20/400) received a single subretinal injection of MA09-hRPE cells, starting at a dose of 50,000 MA09-hRPE cells (three patients), 100,000 MA09-hRPE cells transplanted (three patients), 150,000 MA09-hRPE cells transplanted (three patients) and increasing to a maximum dose of 200,000 MA09-hRPE cells transplanted (one patient). Three patients with severe to moderate vision loss (visual acuity <= 20/100) received a dose of 100,000 MA09-hRPE cells. All patients who participated in the core protocol are eligible for participation in this follow-up protocol.

The first visit of this long term follow-up protocol will correspond to the last visit of the core protocol, and will take place at 12 months post cell implantation. Informed consent will be obtained at this visit.

Patients will be evaluated at 18, 24, 36, 48 and 60 months post-transplant (or more frequently as clinically indicated). Follow-up will include obtaining information about ophthalmological findings and events of special interest as defined in the Primary Outcomes. At the last visit of this follow-up study, whether at 60 months post-transplant or at early discontinuation, patients will be invited to participate in a Safety Surveillance Study for an additional 10 years, under a separate protocol, which will continue to monitor the long term risks of MA09-hRPE cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Must have been treated with hESC-RPE cell transplant in the core protocol.
* Able to understand and willing to sign the informed consent to participate in the follow-up study.

Exclusion Criteria:

* There are no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is by invitation only for previous participants in the core protocol.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Safety assessed by Adverse Events (AEs) of special interest in regards to the investigational product | 4 years
  This will include obtaining information about ophthalmological findings and Serious Adverse Events (SAEs) that are neurologic, infectious, hematologic or fatal, pregnancy in a female subject or the partner of a male subject and pregnancy outcome, any adverse event (AE) that causes a subject to withdraw from the study, any new diagnosis of an ocular or immune-mediated disorder, cancer, ectopic or proliferative cell growth (Retinal pigment epithelium (RPE) or non-RPE) with adverse clinical consequence, and unexpected, clinically significant AEs possibly related to the cell transplant procedure or the investigational product (MA09-hRPE cells).

SECONDARY OUTCOMES:
Incidence of graft failure or rejection | 4 years
  Evidence of graft failure or rejection will consist of: Presence of retinal edema, cystoid macular edema, retinal white dots, retinal hemorrhage, serous retinal detachment, subretinal exudates, subretinal fibrosis, or vascular and/or optic disc leakage, elevated intraocular pressure or hypotony. Evidence of unanticipated and persistent or increasing non-infectious ocular inflammation (e.g., vasculitis, retinitis, choroiditis, vitritis, pars planitis, anterior segment inflammation/uveitis).
Number of patients with changes in ocular examinations or images | 4 years
  The number of patients with clinically significant absolute values or changes from baseline in Intra-ocular pressure (IOP) and Best Corrected Visual Acuity (BCVA) will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Institute for Regenerative Medicine
Locations (3):
- United States (3):
  - Jules Stein Eye Institute, UCLA School of Medicine, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Wills Eye Institute-Mid Atlantic Retina, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Result] Schwartz SD, Hubschman JP, Heilwell G, Franco-Cardenas V, Pan CK, Ostrick RM, Mickunas E, Gay R, Klimanskaya I, Lanza R. Embryonic stem cell trials for macular degeneration: a preliminary report. Lancet. 2012 Feb 25;379(9817):713-20. doi: 10.1016/S0140-6736(12)60028-2. Epub 2012 Jan 24. PMID 22281388
- [Result] Schwartz SD, Regillo CD, Lam BL, Eliott D, Rosenfeld PJ, Gregori NZ, Hubschman JP, Davis JL, Heilwell G, Spirn M, Maguire J, Gay R, Bateman J, Ostrick RM, Morris D, Vincent M, Anglade E, Del Priore LV, Lanza R. Human embryonic stem cell-derived retinal pigment epithelium in patients with age-related macular degeneration and Stargardt's macular dystrophy: follow-up of two open-label phase 1/2 studies. Lancet. 2015 Feb 7;385(9967):509-16. doi: 10.1016/S0140-6736(14)61376-3. Epub 2014 Oct 15. PMID 25458728
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=383